CLINICAL TRIAL: NCT07382921
Title: Efficacy and Safety of Pregabalin/Tizanidine vs. Pregabalin in Patients With Fibromyalgia: a Prospective, Randomized, Open-label, Blinded Endpoint (PROBE) Trial
Brief Title: Efficacy and Safety of Pregabalin/Tizanidine vs. Pregabalin in Patients With Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: People's Hospital of Xinjiang Uygur Autonomous Region (Other); Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-217-03-08
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia; Pregabalin; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin; tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin monotherapy group (Active Comparator)
  Interventions: Drug: Pregabalin
- Pregabalin with tizanidine group (Experimental)
  Interventions: Drug: Pregabalin with tizanidine

INTERVENTIONS:
Drug: Pregabalin — The patients receive open-label pregabalin (Pfizer Pharmaceutical Co. Ltd, New York) titration therapy. In the first week, patients receive the starting dose of 150 mg/day (75 mg twice daily) escalated, based on efficacy and tolerability, at weekly visits to increase by 150 mg per week. A final dose of 450 mg/day (225 mg twice daily). However, during this flexible dose titration, the final dose arrived at during the maximal tolerated dose week (week 3 of the treatment period) could be lower than the ceiling dose of 450 mg, if the patient could not tolerate the dose increase, it is reduce to the pre-escalation dose. Thus, this trial will not use a forced titration to the ceiling dose of 450 mg/day.
  Arms: Pregabalin monotherapy group
Drug: Pregabalin with tizanidine — All patients receive tizanidine in an open-label fashion. The tizanidine dose is slowly escalated over approximately 3 weeks. The initial dosage is 2 mg/d at bedtime. The dosage is increased by 2 mg every 2 days in the first week in 3 divided doses. The dosage is then increased more rapidly by 4 mg every 2 days in the second week divided 3 times a day. During the third week, the dose was further escalated by 6 mg every 2 days to a maximum of 24 mg/d divided 3 times a day. If a patient could not tolerate a particular current specific dosage increase because of side effects, he or she is maintain at the previous dosage during the trial period. The patients receive open-label pregabalin (Pfizer Pharmaceutical Co. Ltd, New York) titration therapy. In the first week, patients receive the starting dose of 150 mg/day (75 mg twice daily) escalated, based on efficacy and tolerability, at weekly visits to increase by 150 mg per week. A final dose of 450 mg/day (225 mg twice daily).
  Arms: Pregabalin with tizanidine group

SUMMARY:
Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread pain, fatigue, and emotional disorders. Its onset is related to factors such as central sensitization and imbalance of neurotransmitters. The current mainstream treatments include pregabalin, but the efficacy of pregabalin is limited, with only 25%-40% pain relief rate, and adverse reactions are common.Tizanidine is an imidazoline derivative and a centrally acting alpha-2 receptor agonist with skeletal muscle relaxant, sedative and anxiolytic properties.we carried out an open-label clinical trial in order to evaluate the efficacy and safety of combined treatment with tizanidine and pregabalin for pain in FM.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 18-65 years. 2.Fulfill the 2016 updated American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia.

  3.Sufficient cognitive function, visual acuity and language skills to complete questionnaires and pain diaries and to participate in telephone communication with study nurses to permit titration of the study drugs.

  4.Experienced daily pain (≥4/10 on a numerical rating scale) for at least 3 months.

Exclusion Criteria:

* 1.Presence of a painful condition, including inflammatory rheumatic disease, more than 50% as severe as but distinct from fibromyalgia.

  2.Women who are pregnant or lactating. 3.Women of childbearing potential not using adequate contraceptives. 4.End-stage kidney or liver disease. 5.Unstable cardiovascular disease (myocardial infarction within the preceding year, unstable angina, or congestive heart failure) or clinically relevant abnormal 12-lead electrocardiogram.

  6.Any poorly controlled medical condition that, in the opinion of the investigator, would interfere with proper conduct of the trial.

  7.Severe depression, as determined by a Beck Depression Inventory-II score of 29 or more suicidal ideation, as determined by a Beck Depression Inventory-II item 9 score of 2 or more any current major psychiatric disorder (e.g., schizophrenia, bipolar disorder) that is not well controlled.

  8.Hypersensitivity to any of the study medications. 9.Any current alcohol or drug abuse or dependence (except nicotine and caffeine).

  10.Those taking more than 90 mg morphine equivalents per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Average pain intensity | baseline , 12 weeks
  The primary outcome is change from baseline to 12 weeks of treatment in average pain intensity during the last 7 days on an 11-point rating scale (ranging from 0 = "no pain" to 10 = "unbearable pain") using the first item from the symptom part of the Fibromyalgia Impact Questionnaire Revised (FIQR)

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised | weekly(from baseline to 24 weeks)
  The FIQR is a well-validated multidimensional instrument that measures participant-rated overall severity of fibromyalgia, including intensity of pain, physical function, fatigue, morning tiredness, depression, anxiety, job difficulty, and overall well-being. Each item is standardized on a scale ranging from 0 to 10, with lower scores indicating more improvement or less negative impact. In addition, FIQR is also assessed weekly during the intervention period for all groups of participants as well as at the 24-week time points as secondary outcomes.
Medical Outcome Study Short Form 36 Health Survey (SF-36) | baseline , 4, 8, 12, 16, 20, and 24 weeks
  Health Related Quality of Life assessments are made using the Medical Outcome Study Short Form 36 Health Survey (SF-36). The SF-36 is a self-administered, 36-item questionnaire that assesses the concepts of physical functioning, role limitations due to physical problems, social function, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. Summary scores include physical function, mental function, and combined total function. Scores range from 0 to 100, with higher scores indicating better health status.
The Patient's Global Assessment | baseline , 4, 8, 12, 16, 20, and 24 weeks
  The Patient's Global Assessment (Global Visual Analogue Scale) is a visual analogue scale that measures the level of fibromyalgia severity on a 10-point scale with 10 reflecting the most extreme severity and 0 reflecting no severity.
The Beck II Depression Inventory | baseline , 4, 8, 12, 16, 20, and 24 weeks
  The Beck II Depression Inventory (BDI) is a 21-question, validated, self-report instrument that measures the severity of depressive symptoms (each scored 0-3, sum=0-63). Higher scores reflect a greater degree of symptom severity. The total questionnaire score ranges from 0 to 63 points. The result is interpreted by the usual classifications as follows: no depression (0-9 points), mild depression (10-18 points), moderate depression (19-29 points) and severe depression (>30 points).
The Pittsburgh Sleep Quality Index | baseline , 4, 8, 12, 16, 20, and 24 weeks
  The Pittsburgh Sleep Quality Index is an 11-item, validated, self-report questionnaire that measures sleep quality. Lower scores are associated with better sleep quality. This questionnaire has 7 dimensions: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction. Each dimension is scored from 0 (no problems) to 3 (severe problems), where the total score varies in a range from 0 to 21 points.
The Hospital Anxiety and Depression Scale | baseline , 4, 8, 12, 16, 20, and 24 weeks
  The Hospital Anxiety and Depression Scale is a 14-item, validated, self-report questionnaire that assesses levels of depression and anxiety. Higher scores reflect greater levels of anxiety and depression.
The Perceived Stress Scale | baseline , 4, 8, 12, 16, 20, and 24 weeks
  The Perceived Stress Scale is the most widely used psychological instrument for measuring the perception of stress. The 10-item scale also includes a number of direct queries about current levels of experienced stress. For this instrument, higher scores reflect a greater degree of symptom severity.
Pain distribution | baseline , 4, 8, 12, 16, 20, and 24 weeks
  Pain distribution: assessed by the Widespread Pain Index (WPI) from the 2016 diagnostic criteria for fibromyalgia.
Frequency and severity of AEs | baseline , 4, 8, 12, 16, 20, and 24 weeks
  Frequency and severity of AEs, Patient safety will be ensured by vigilant AE assessment and judicious drug titration. Any occurrences of major AEs will be tracked as secondary outcomes and also reported to the Ethics Board. Assessment and reporting of AEs will adhere to Consolidated Standards for Reporting Trials recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University in Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.